CLINICAL TRIAL: NCT06104540
Title: Comparison of the Effects of Liquid Vaseline and Olive Oil on Itching and Scarring in Scald Burns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Nuray Çetintaş, Principal investigator, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AYBUSBENURAYCETINTAS0000000001
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Scald Burn; Itching; Hypertrophic Scarring
Keywords: scald burns; nursing care; oliveoil; liquid vaseline; itching; hypertrophic scarring
MeSH Terms: conditions — Pruritus; Cicatrix, Hypertrophic

STUDY DESIGN:
Intervention Model Description: A preliminary study will be conducted with 24 patients, 8 in the control group and 8 in the experimental group I olive oil and the experimental group II 8 with liquid vaseline. Patients will be divided into control and experimental groups by simple stratified randomization method.
  In order to prevent the choice of treatment from being at the discretion of the investigator, it is necessary to ensure that the patients are randomly assigned to the study groups. The easiest method for this is simple randomization. The envelope drawing method will be used for randomization and patients who meet the research criteria will be stratified according to gender. To ensure gender stratification in the control and experimental groups, male patients will be assigned to control and experimental groups and female patients will be assigned to control and experimental groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental I Liquid Vaseline (Experimental): Liquid vaseline will be applied to the Experimental I group twice a day according to the oil application protocol
  Interventions: Other: Experimental I liquid vaseline groups
- Experimental II Extra Virgin Olive Oil (Experimental): Extra Virgin Olive Oil will be applied to the Experimental I group twice a day according to the oil application protocol
  Interventions: Other: Experimental II extra virgin olive oil groups
- Control group (Experimental): No application will be made to the control group other than the institution's recommendations.
  Interventions: Other: Control Croup

INTERVENTIONS:
Other: Experimental I liquid vaseline groups — Patients in the liquid vaseline group will apply liquid vaseline twice a day for 3 months. Depending on the size of the burn area, 5-10 ml of liquid petroleum jelly will be applied to the burn area by massaging for 5 minutes twice a day, and each application will be recorded in the application follow-up form. Patients will be visited on the 15th day, first month, second month, and third month after the application begins.
  Arms: Experimental I Liquid Vaseline
Other: Experimental II extra virgin olive oil groups — Patients in the extra virgin olive oil group will apply extra virgin olive oil twice a day for 3 months. Depending on the size of the burn area, 5-10 ml of liquid petroleum jelly will be applied to the burn area by massaging for 5 minutes twice a day, and each application will be recorded in the application follow-up form. Patients will be visited on the 15th day, first month, second month, and third month after the application begins.
  Arms: Experimental II Extra Virgin Olive Oil
Other: Control Croup — No intervention will be made other than the recommendations of the institution's physicians and nurses.
  Arms: Control group

SUMMARY:
Pain, itching, hypertrophic scar formation after wound healing in burn patients complications, sleep disturbances in patients, anxiety, depression, and daily life It may disrupt activities and deterioration in quality of life. Liquid petroleum jelly and olive oil have no side effects, moisturizing properties, or wound-healing treatment of burns due to their positive effects on symptoms such as itching. can be used to alleviate burns. The project found the use of liquid petroleum jelly and olive oil to determine the effect on itching and scarring in burn patients. After burns reduction of symptoms such as itching, dryness, hypertrophic scarring, and patient comfort. Provision of care is a part of nursing care. In studies, itching and scarring there is insufficient evidence regarding the treatment methods applied for its treatment is observed. In addition, the effect of olive oil and liquid petroleum jelly on itching and scarring no scientific study was found. The results of the project were found to be significant in terms of post-burn itching providing evidence of hypertrophic scar management and contributing to ongoing studies is expected to be found. Since there are no similar studies in the literature, a preliminary study with 24 patient applications will be made. In line with the data obtained from the pre-application, the sample calculation will be made and the application will continue by making the necessary arrangements. Patients will be divided into experimental and control groups by simple randomization. All patient groups individual data collection forms on the first day; 12 individual data collection forms on the first day, 15th day, first, second, and third months Itemized Itch Severity Scale, Patient and Observer Scar Scale to be applied in Burn Patients and the wound area will be photographed. Patients in the control group will be given no application will be made. Liquid petroleum jelly and olive oil group before the study training will be given and they will massage the recommended product twice a day for 3 months and will be asked to record them. The data obtained at the end of the project will be statistically analyzed and results will be presented.

DETAILED DESCRIPTION:
In addition to localized damage, burn is defined as a comprehensive trauma that affects the whole organism and determines the prognosis with its physiological response and can cause physical, psychological, sociological, and economic problems in the individual. Although the etiology of burn injuries varies according to industrialization, socioeconomic, cultural, educational, and age groups, scald burns, flame burns, and electrical burns are the most common causes of burn injuries. Esen et al. (2021) reported that scald burns ranked first among the causes of burns with 37.2% in their study. Although survival in patients has increased with advances in burn treatment, wound healing, and understanding of scar pathophysiology, burns are still an important cause of morbidity. In these patients, postburn pruritus and hypertrophic scarring is a common and important complication that occurs during the wound-healing process Histamine produced by mast cells during the injury process plays a role in the development of post-burn itching and acute itching begins with wound closure. The prevalence of itching after burns is reported to be 80-100% The risk of itching increases in patients with large burn surface area, surgical procedures related to burn, hypertrophic scarring, female gender, dry skin, limb, and facial burns In addition to itching, patients may experience various sensory disturbances such as "pinprick", stabbing, or burning after burns.

Another problem affecting patients after burns is the development of hypertrophic scarring. Abnormal increase of collagen and glycoprotein and transepidermal water loss during the wound healing process can cause hypertrophic scarring or keloid. In wound healing, hypertrophic scarring occurs within four weeks after complete reepithelialization and regresses in approximately 15 months. The incidence of hypertrophic scar formation following burn injuries ranges from 34% to 94%. In one study, itching, pain, and paresthesia requiring treatment were observed in patients with hypertrophic scarring, and it is recommended to identify and prevent risk factors for treatment and symptom control.

Alleviation of itching symptoms after burns and early diagnosis of hypertrophic scar development is important in rehabilitation. Itching and hypertrophic scarring can cause cosmetic problems, severe functional disability, pain, sleep disorders, re-damage of fragile skin, and risk of infection with microorganism colonization, anxiety, and depression. Topical moisturizers, cold application, pressure garments, antihistamines, massage, psychological therapy and dermatological treatments, surgical techniques, and laser treatment can be applied in the treatment. The effectiveness of all these treatment methods is limited and there is insufficient evidence.

One of the factors that make scars visible is dry skin due to transepidermal water loss and skin should be kept moist to minimize the appearance of scars. The use of moisturizers has been identified as one of the components of treatment to reduce itching and hypertrophic scarring. Moisturizers are available in the form of plant extracts and various oils. Various topical products with moisturizing properties such as olive oil, and St. John's wort can be used in the treatment of burns and alleviation of itching and dryness symptoms after burns due to their cheap and easy availability, lack of side effects, moisturizing properties, positive properties on wound healing. Olive oil contains fatty components such as oleic acid, phenolic compounds, chlorophyll, and vitamin E. These components accelerate wound healing, moisturize the skin, and provide elasticity to the skin. In the study investigating the effect of olive oil and flaxseed on burn healing, it was shown that when the oils were applied as a mixture, they reduced inflammation and had a positive effect on wound size.

One of the products used for moisturizing is liquid petroleum jelly. Liquid petroleum jelly is obtained from liquid petroleum consisting of colorless, odorless, oily saturated hydrocarbons. It is widely used for cosmetic purposes and is included in the composition of many topical products. It reduces skin water loss, moisturizes the skin, reduces itching symptoms, acts as a barrier, and protects skin integrity. Wang et al. (2020) found that liquid petroleum jelly was more effective in wound healing and prevention of infection compared to normal saline in their research evaluating the effectiveness of liquid petroleum jelly in the treatment of burn wounds.

Problems such as itching, dryness, scarring, and hypertrophic scarring after burns negatively affect the patient's quality of life and body image. Therefore, the nurse should know the treatment and preventive measures and evaluate the effectiveness of the interventions using appropriate measurement tools. It is stated in the literature that the substances in the composition of olive oil support wound healing and moisturizing properties, but there are no clinical studies investigating the effect of olive oil and liquid petroleum jelly on itching and scarring in burn wounds. This study aims to determine the effect of topically applied olive oil and liquid petroleum jelly on itching and scarring in post-burn patients.

Expected benefits and risks of research, The study will be conducted to determine the effect of olive oil and liquid petroleum jelly on itching and scarring that occur during the healing period after a scald burn.

This study aims to help patients cope with itching and scarring problems that occur in the post-burn period and to shed light on the nursing interventions to be made for a more qualified life.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65,
* With a total body burn area of less than 15% 2nd degree scald burn,
* Wwhose treatment has been completed and who do not need dressing and do not have open wounds,
* Who do not have any allergies,
* Who can read and write,
* Who do not have cognitive problems,
* Who do not have communication problems,
* Who live in Ankara and who volunteer to participate in the study.

Exclusion Criteria:

* Patients with burns on the face and neck,
* Ppatients with dermatologic diseases and patients using antihistamines will not be included.
* Patients who do not want to continue the study,
* Who develop an allergic reaction during the follow-up period,
* Who start treatment during the follow-up period due to itching,
* Wwho have not applied more than 20% liquid vaseline/olive oil during the 3-month follow-up period (60 applications/30 days; more than 36 applications out of 180 applications) will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
12-item itch scale scores | Before you start applying liquid vaseline
  assessment of itching severity. The lowest score on the scale is 3, indicating minimum itching, while the lowest score on the scale is 3.
  The high score of 22 points indicates severe itching. Scale scores It is assumed that as the score increases, the patient's level of exposure to itching increases.
Observer scar assesment scale score | Before you start applying liquid vaseline
  assessment of hypertrophic scar.Observer Scar Assessment Scale, Each item is scored on a Likert-type scale between 1 and 10. has. 1 indicates "normal skin" and 10 indicates "worst scar evaluation". The lowest score a patient can get on the scale is 6, indicating normal skin and the highest score is 60.
  It represents the worst scar imaginable.
12-item itch scale scores | Before you start applying extra virgin olive oil
  assessment of itching severity. The lowest score on the scale is 3, indicating minimum itching, while the lowest score on the scale is 3.
  The high score of 22 points indicates severe itching. Scale scores It is assumed that as the score increases, the patient's level of exposure to itching increases.
Patient scar assesment scale score | Before you start applying extra virgin olive oil
  assessment of hypertrophic scar. Patient Scar Assessment Scale, 1 being "normal skin", 10 being "worst scar".
  shows the evaluation. The lowest score a patient can get on the scale is 6, Normal skin, the highest score of 60, the worst imaginable scar, The scale score is calculated based on the first 6 items. The general opinion about scar The 7th item, which questions questions, has only scoring criteria and is evaluated.
Observer scar assesment scale score | Before you start applying extra virgin olive oil
  assessment of hypertrophic scar. Observer Scar Assessment Scale, Each item is scored on a Likert-type scale between 1 and 10. has. 1 indicates "normal skin" and 10 indicates "worst scar evaluation". The lowest score a patient can get on the scale is 6, indicating normal skin and the highest score is 60.
  It represents the worst scar imaginable.
12-item itch scale scores | will be applied to the control group on the first day
  assessment of itching severity. The lowest score on the scale is 3, indicating minimum itching, while the lowest score on the scale is 3.
  The high score of 22 points indicates severe itching. Scale scores It is assumed that as the score increases, the patient's level of exposure to itching increases.
  Assessment Scale, scar evaluation (vascularization, pigmentation, thickness, irregularity, elasticity, surface area) and scar A total of 7 articles, including 1 article evaluating the general opinion about is formed. Each item is scored on a Likert-type scale between 1 and 10. has. 1 indicates "normal skin" and 10 indicates "worst scar evaluation". The lowest score a patient can get on the scale is 6, indicating normal skin, and the highest score is 60.
  It represents the worst scar imaginable, and the scale score is based on the first 6 items.
  was being calculated
Patient scar assessment scale score | will be applied to the control group on the first day
  assessment of hypertrophic scar. Patient Scar Assessment Scale, 1 being "normal skin", 10 being "worst scar". shows the evaluation. The lowest score a patient can get on the scale is 6, Normal skin, the highest score of 60, the worst imaginable scar, The scale score is calculated based on the first 6 items. The general opinion about scar The 7th item, which questions questions, has only scoring criteria and is evaluated.
Observer scar assesment scale score | will be applied to the control group on the first day
  assessment of hypertrophic scar. Observer Scar Assessment Scale, each item is scored on a Likert-type scale between 1 and 10.
  has. 1 indicates "normal skin" and 10 indicates "worst scar evaluation". The lowest score a patient can get on the scale is 6, indicating normal skin, and the highest score is 60.
  It represents the worst scar imaginable.
Patient scar assesment scale score | Before you start applying liquid vaseline
  assessment of hypertrophic scar. Patient Scar Assessment Scale, 1 being "normal skin", 10 being "worst scar".
  shows the evaluation. The lowest score a patient can get on the scale is 6, Normal skin, the highest score of 60, the worst imaginable scar, The scale score is calculated based on the first 6 items. The general opinion about scar The 7th item, which questions questions, has only scoring criteria and is evaluated.

SECONDARY OUTCOMES:
12-item itch scale scores | 15 days after starting liquid vaseline application
  assessment of itching severity. The lowest score on the scale is 3, indicating minimum itching, while the lowest score on the scale is 3.
  The high score of 22 points indicates severe itching. Scale scores It is assumed that as the score increases, the patient's level of exposure to itching increases.
Patient scar assesment scale score | 15 days after starting liquid vaseline application
  assessment of hypertrophic scar. Patient Scar Assessment Scale, 1 being "normal skin", 10 being "worst scar". shows the evaluation. The lowest score a patient can get on the scale is 6, Normal skin, the highest score of 60, the worst imaginable scar, The scale score is calculated based on the first 6 items. The general opinion about scar The 7th item, which questions questions, has only scoring criteria and is evaluated.
Observer scar assesment scale score | 15 days after starting liquid vaseline application
  assessment of hypertrophic scar. Observer Scar Assessment Scale, each item is scored on a Likert-type scale between 1 and 10.
  has. 1 indicates "normal skin" and 10 indicates "worst scar evaluation". The lowest score a patient can get on the scale is 6, indicating normal skin and the highest score is 60.
  It represents the worst scar imaginable.
12-item itch scale scores | 15 days after starting extra virgin olive oil
  assessment of itching severity. The lowest score on the scale is 3, indicating minimum itching, while the lowest score on the scale is 3.
  The high score of 22 points indicates severe itching. Scale scores It is assumed that as the score increases, the patient's level of exposure to itching increases.
Patient scar assesment scale score | 15 days after starting extra virgin olive oil
  assessment of hypertrophic scar. Patient Scar Assessment Scale, 1 being "normal skin", 10 being "worst scar". shows the evaluation. The lowest score a patient can get on the scale is 6, Normal skin, the highest score of 60, the worst imaginable scar, The scale score is calculated based on the first 6 items. The general opinion about scar The 7th item, which questions questions, has only scoring criteria and is evaluated.
Observer scar assessment scale score | 15 days after starting extra virgin olive oil
  assessment of hypertrophic scar. Observer Scar Assessment Scale, each item is scored on a Likert-type scale between 1 and 10.
  has. 1 indicates "normal skin" and 10 indicates "worst scar evaluation". The lowest score a patient can get on the scale is 6, indicating normal skin and the highest score is 60.
  It represents the worst scar imaginable.
12-item itch scale scores | control group will be applied on the 15th day
  assessment of itching severity. The lowest score on the scale is 3, indicating minimum itching, while the lowest score on the scale is 3.
  The high score of 22 points indicates severe itching. Scale scores It is assumed that as the score increases, the patient's level of exposure to itching increases
Patient scar assessment scale score | control group will be applied on the 15th day
  assessment of hypertrophic scar. Patient Scar Assessment Scale, 1 being "normal skin", 10 being "worst scar". shows the evaluation. The lowest score a patient can get on the scale is 6, Normal skin, the highest score of 60, the worst imaginable scar, The scale score is calculated based on the first 6 items. The general opinion about scar The 7th item, which questions questions, has only scoring criteria and is evaluated.
Observer scar assessment scale score | control group will be applied on the 15th day
  assessment of hypertrophic scar. Observer Scar Assessment Scale, each item is scored on a Likert-type scale between 1 and 10.
  has. 1 indicates "normal skin" and 10 indicates "worst scar evaluation". The lowest score a patient can get on the scale is 6, indicating normal skin and the highest score is 60.
  It represents the worst scar imaginable.

OTHER OUTCOMES:
12-item itch scale scores | One month after starting liquid vaseline application
  assessment of itching severity. The lowest score on the scale is 3, indicating minimum itching, while the lowest score on the scale is 3.
  The high score of 22 points indicates severe itching. Scale scores It is assumed that as the score increases, the patient's level of exposure to itching increases.
Patient scar assessment scale score | One month after starting liquid vaseline application
  assessment of hypertrophic scar. Patient Scar Assessment Scale, 1 being "normal skin", 10 being "worst scar". shows the evaluation. The lowest score a patient can get on the scale is 6, Normal skin, the highest score of 60, the worst imaginable scar, The scale score is calculated based on the first 6 items. The general opinion about scar The 7th item, which questions questions, has only scoring criteria and is evaluated.
Observer scar assessment scale score | One month after starting liquid vaseline application
  assessment of hypertrophic scar. Observer Scar Assessment Scale, each item is scored on a Likert-type scale between 1 and 10.
  has. 1 indicates "normal skin" and 10 indicates "worst scar evaluation". The lowest score a patient can get on the scale is 6, indicating normal skin and the highest score is 60.
  It represents the worst scar imaginable.
12-item itch scale scores | One month after starting extra virgin olive oil application
  assessment of itching severity. The lowest score on the scale is 3, indicating minimum itching, while the lowest score on the scale is 3.
  The high score of 22 points indicates severe itching. Scale scores It is assumed that as the score increases, the patient's level of exposure to itching increases.
Patient scar assesment scale score | One month after starting extra virgin olive oil application
  assessment of hypertrophic scar. Patient scar assessment scale,1 being "normal skin", 10 being "worst scar".
  shows the evaluation. The lowest score a patient can get from the scale is 6, Normal skin, the highest score of 60, the worst imaginable scar, The scale score is calculated based on the first 6 items. General opinion about scar The 7th item, which questions questions, has only scoring criteria and is evaluated.
Observer scar assesment scale score | One month after starting extra virgin olive oil
  assessment of hypertrophic scar. Observer Scar Assessment Scale, each item is scored on a Likert-type scale between 1 and 10.
  has. 1 indicates "normal skin" and 10 indicates "worst scar evaluation". The lowest score a patient can get on the scale is 6, indicating normal skin and the highest score is 60.
  It represents the worst scar imaginable.
12-item itch scale scores | control group will be applied in the first month
  assessment of itching severity. The lowest score on the scale is 3, indicating minimum itching, while the lowest score on the scale is 3.
  The high score of 22 points indicates severe itching. Scale scores It is assumed that as the score increases, the patient's level of exposure to itching increases.
Patient scar assesment scale score | control group will be applied in the first month
  assessment of hypertrophic scar. Patient Scar Assessment Scale, 1 being "normal skin", 10 being "worst scar". shows the evaluation. The lowest score a patient can get on the scale is 6, Normal skin, the highest score of 60, the worst imaginable scar, The scale score is calculated based on the first 6 items. The general opinion about scar The 7th item, which questions questions, has only scoring criteria and is evaluated.
Observer scar assesment scale score | control group will be applied in the first month
  assessment of hypertrophic scar. Observer Scar Scale, each item is scored on a Likert-type scale between 1 and 10.
  has. 1 indicates "normal skin" and 10 indicates "worst scar evaluation". The lowest score a patient can get on the scale is 6, indicating normal skin and the highest score is 60.
  It represents the worst scar imaginable.
12-item itch scale scores | Two month after starting liquid vaseline application
  assessment of itching severity. The lowest score on the scale is 3, indicating minimum itching, while the lowest score on the scale is 3.
  The high score of 22 points indicates severe itching. Scale scores It is assumed that as the score increases, the patient's level of exposure to itching increases.
Patient scar assesment scale score | Two month after starting liquid vaseline application
  assessment of hypertrophic scar. Patient scar assessment scale,1 being "normal skin", and 10 being "worst scar".
  shows the evaluation. The lowest score a patient can get on the scale is 6, Normal skin, the highest score of 60, the worst imaginable scar, The scale score is calculated based on the first 6 items. The general opinion about scar The 7th item, which questions questions, has only scoring criteria and is evaluated.
Observer scar assesment scale score | Two month after starting liquid vaseline application
  assessment of hypertrophic scar. Observer Scar Scale, each item is scored on a Likert-type scale between 1 and 10.
  has. 1 indicates "normal skin" and 10 indicates "worst scar evaluation". The lowest score a patient can get on the scale is 6, indicating normal skin and the highest score is 60.
  It represents the worst scar imaginable.
12-item itch scale scores | Two month after starting extra virgin olive oil application
  assessment of itching severity. The lowest score on the scale is 3, indicating minimum itching, while the lowest score on the scale is 3.
  The high score of 22 points indicates severe itching. Scale scores It is assumed that as the score increases, the patient's level of exposure to itching increases.
Patient scar assesment scale score | Two month after starting extra virgin olive oil application
  assessment of hypertrophic scar. Patient Scar Assessment Scale, 1 being "normal skin", 10 being "worst scar". shows the evaluation. The lowest score a patient can get on the scale is 6, Normal skin, the highest score of 60, the worst imaginable scar, The scale score is calculated based on the first 6 items. The general opinion about scar The 7th item, which questions questions, has only scoring criteria and is evaluated.
Observer scar assesment scale score | Two month after starting extra virgin olive oil application
  assessment of hypertrophic scar. Observer Scar Scale, each item is scored on a Likert-type scale between 1 and 10.
  has. 1 indicates "normal skin" and 10 indicates "worst scar evaluation". The lowest score a patient can get on the scale is 6, indicating normal skin and the highest score is 60.
  It represents the worst scar imaginable.
12-item itch scale scores | The control group will be applied in the second month
  assessment of itching severity. The lowest score on the scale is 3, indicating minimum itching, while the lowest score on the scale is 3.
  The high score of 22 points indicates severe itching. Scale scores It is assumed that as the score increases, the patient's level of exposure to itching increases.
Patient scar assesment scale score | The control group will be applied in the second month
  assessment of hypertrophic scar. Patient scar assessment scale, 1 being "normal skin", and 10 being "worst scar".
  shows the evaluation. The lowest score a patient can get on the scale is 6, Normal skin, the highest score of 60, the worst imaginable scar, The scale score is calculated based on the first 6 items. The general opinion about scar The 7th item, which questions questions, has only scoring criteria and is evaluated.
Observer scar assesment scale score | The control group will be applied in the second month
  assessment of hypertrophic scar. Observer Scar Scale, each item is scored on a Likert-type scale between 1 and 10.
  has. 1 indicates "normal skin" and 10 indicates "worst scar evaluation". The lowest score a patient can get on the scale is 6, indicating normal skin and the highest score is 60.
  It represents the worst scar imaginable.
12-item itch scale scores | Three month after starting liquid vaseline application
  assessment of itching severity. The lowest score on the scale is 3, indicating minimum itching, while the lowest score on the scale is 3.
  The high score of 22 points indicates severe itching. Scale scores It is assumed that as the score increases, the patient's level of exposure to itching increases.
Patient scar assesment scale score | Three month after starting liquid vaseline application
  assessment of hypertrophic scar. Patient Scar Assessment Scale, 1 being "normal skin", 10 being "worst scar". shows the evaluation. The lowest score a patient can get from the scale is 6, Normal skin, the highest score of 60, the worst imaginable scar, The scale score is calculated based on the first 6 items. General opinion about scar The 7th item, which questions questions, has only scoring criteria and is evaluated.
Oobserver scar assesment scale score | Three month after starting liquid vaseline application
  assessment of hypertrophic scar. Observer Scar Scale, each item is scored on a Likert-type scale between 1 and 10.
  has. 1 indicates "normal skin" and 10 indicates "worst scar evaluation". The lowest score a patient can get on the scale is 6, indicating normal skin and the highest score is 60.
  It represents the worst scar imaginable.
12-item itch scale scores | Three month after starting extra virgin olive oil application
  assessment of itching severity. The lowest score on the scale is 3, indicating minimum itching, while the lowest score on the scale is 3.
  The high score of 22 points indicates severe itching. Scale scores It is assumed that as the score increases, the patient's level of exposure to itching increases.
Patient scar assesment scale score | Three month after starting extra virgin olive oil application
  assessment of hypertrophic scar. Patient Scar Assessment Scale, 1 being "normal skin", 10 being "worst scar". shows the evaluation. The lowest score a patient can get from the scale is 6, Normal skin, the highest score of 60, the worst imaginable scar, The scale score is calculated based on the first 6 items. General opinion about scar The 7th item, which questions questions, has only scoring criteria and is evaluated.
Observer scar assesment scale score | Three month after starting extra virgin olive oil application
  assessment of hypertrophic scar. Observer Scar Scale, each item is scored on a Likert-type scale between 1 and 10.
  has. 1 indicates "normal skin" and 10 indicates "worst scar evaluation". The lowest score a patient can get on the scale is 6, indicating normal skin and the highest score is 60.
  It represents the worst scar imaginable.
12-item itch scale scores | The control group will be applied in the third month
  assessment of itching severity. The lowest score on the scale is 3, indicating minimum itching, while the lowest score on the scale is 3.
  The high score of 22 points indicates severe itching. Scale scores It is assumed that as the score increases, the patient's level of exposure to itching increases.
Patient scar assesment scale score | The control group will be applied in the third month
  assessment of hypertrophic scar. Patient Scar Assessment Scale, 1 being "normal skin", 10 being "worst scar". shows the evaluation. The lowest score a patient can get on the scale is 6, Normal skin, the highest score of 60, the worst imaginable scar, The scale score is calculated based on the first 6 items. The general opinion about scar The 7th item, which questions questions, has only scoring criteria and is evaluated.
Observer scar assesment scale score | The control group will be applied in the third month
  assessment of hypertrophic scar. Observer Scar Scale, each item is scored on a Likert-type scale between 1 and 10.
  has. 1 indicates "normal skin" and 10 indicates "worst scar evaluation". The lowest score a patient can get on the scale is 6, indicating normal skin and the highest score is 60.
  It represents the worst scar imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Merve AKIN, Ass Prof, Principal Investigator — Ankara City Hospital Bilkent; Nuray Çetintaş, Master, Principal Investigator; Sema Koçaşlı, Prof Asst Dr, Study Director
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is planned to share all IPD datasets collected according to the results of the pre-implementation.

REFERENCES:
- [Background] Xiao Y, Sun Y, Zhu B, Wang K, Liang P, Liu W, Fu J, Zheng S, Xiao S, Xia Z. Risk factors for hypertrophic burn scar pain, pruritus, and paresthesia development. Wound Repair Regen. 2018 Mar;26(2):172-181. doi: 10.1111/wrr.12637. PMID 29719102
- [Background] Wang JJ, Yang L, Chen X. [Observation on the effect of liquid paraffin as adjuvant therapy in treating residual wounds of patients with severe burns]. Zhonghua Shao Shang Za Zhi. 2020 Apr 20;36(4):304-307. doi: 10.3760/cma.j.cn501120-20190316-00122. Chinese. PMID 32340421
- [Background] Vercelli S, Ferriero G, Sartorio F, Stissi V, Franchignoni F. How to assess postsurgical scars: a review of outcome measures. Disabil Rehabil. 2009;31(25):2055-63. doi: 10.3109/09638280902874196. PMID 19888834
- [Background] Sharif F, Crushell E, O'Driscoll K, Bourke B. Liquid paraffin: a reappraisal of its role in the treatment of constipation. Arch Dis Child. 2001 Aug;85(2):121-4. doi: 10.1136/adc.85.2.121. No abstract available. PMID 11466186
- [Background] Reich A, Bozek A, Janiszewska K, Szepietowski JC. 12-Item Pruritus Severity Scale: Development and Validation of New Itch Severity Questionnaire. Biomed Res Int. 2017;2017:3896423. doi: 10.1155/2017/3896423. Epub 2017 Oct 2. PMID 29098154
- [Background] Parnell LK, Nedelec B, Rachelska G, LaSalle L. Assessment of pruritus characteristics and impact on burn survivors. J Burn Care Res. 2012 May-Jun;33(3):407-18. doi: 10.1097/BCR.0b013e318239d206. PMID 22210065
- [Background] Nedelec B, Rachelska G, Parnell LK, LaSalle L. Double-blind, randomized, pilot study assessing the resolution of postburn pruritus. J Burn Care Res. 2012 May-Jun;33(3):398-406. doi: 10.1097/BCR.0b013e318233592e. PMID 21979845
- [Background] Lewis PA, Wright K, Webster A, Steer M, Rudd M, Doubrovsky A, Gardner G. A randomized controlled pilot study comparing aqueous cream with a beeswax and herbal oil cream in the provision of relief from postburn pruritus. J Burn Care Res. 2012 Jul-Aug;33(4):e195-200. doi: 10.1097/BCR.0b013e31825042e2. PMID 22665131
- [Background] Karakoc IB, Ekici B. Maintaining Skin Integrity in Neonates with Sunflower Seed Oil and Liquid Vaseline: A Prospective Randomized Controlled Study. Adv Skin Wound Care. 2022 Dec 1;35(12):1-8. doi: 10.1097/01.ASW.0000891080.13305.75. PMID 36409190
- [Background] Ghanbari A, Masoumi S, Kazemnezhad Leyli E, Mahdavi-Roshan M, Mobayen M. Effects of Flaxseed Oil and Olive Oil on Markers of Inflammation and Wound Healing in Burn Patients: A Randomized Clinical Trial. Bull Emerg Trauma. 2023;11(1):32-40. doi: 10.30476/BEAT.2022.97070.1399. PMID 36818058
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] Chung BY, Kim HB, Jung MJ, Kang SY, Kwak IS, Park CW, Kim HO. Post-Burn Pruritus. Int J Mol Sci. 2020 May 29;21(11):3880. doi: 10.3390/ijms21113880. PMID 32485929
- [Background] Carrougher GJ, Martinez EM, McMullen KS, Fauerbach JA, Holavanahalli RK, Herndon DN, Wiechman SA, Engrav LH, Gibran NS. Pruritus in adult burn survivors: postburn prevalence and risk factors associated with increased intensity. J Burn Care Res. 2013 Jan-Feb;34(1):94-101. doi: 10.1097/BCR.0b013e3182644c25. PMID 23079565
- See also: scholar.google.com.tr — https://turkjdermatol.com/